CLINICAL TRIAL: NCT03926598
Title: User Evaluation of the Guide To Goals Application - a Care Coordination Tool to Translate ADA Clinical Standards of Care for Children With T2D Into Practice
Brief Title: Guide To Goals: A Novel Care Coordination Tool for Children With Type Two Diabetes (T2D)
Acronym: GTG
Status: Completed | Type: Observational
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Emory University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: H18426; P30DK111024 (NIH)
Record Dates: First submitted 2019-04-10; First posted 2019-04-24 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Observational; Mobile Applications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Patients/Caretakers Group: Patients with Type II Diabetes and caretakers of patients with Type II Diabetes.
  Interventions: Behavioral: Patient and/or Family Member Intervention
- Certified Diabetes Educators Group: Diabetes educators who help patients manage their Type II Diabetes.
  Interventions: Behavioral: Certified Diabetes Educator Intervention
- Physician Group: Physicians who help patients manage their Type II Diabetes.
  Interventions: Behavioral: Physician Intervention
- Front Desk Staff: Front desk staff who work with physicians that treat Type II Diabetes.
  Interventions: Behavioral: Front Desk Staff Intervention
- Nurses: Nurses who help patients manage their Type II Diabetes.
  Interventions: Behavioral: Nurse Intervention

INTERVENTIONS:
Behavioral: Patient and/or Family Member Intervention — On the Patient Login Screen, log in using your last name and session ID provided by the research team on the Surveys Screen, click on a pending survey when the survey opens, respond to the survey submit the survey log out of the Guide-Goals Application.
  Groups: Patients/Caretakers Group
Behavioral: Certified Diabetes Educator Intervention — On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen, choose patient Will Owens on the Visit Status Screen, add comments needs to be followed up regarding ketosis education in the comments for provider text box on the Visit Status Screen, add a goal for the patient log out of Goals-to-Guide application.
  Groups: Certified Diabetes Educators Group
Behavioral: Physician Intervention — On the Provider Login Screen, log in using the username and password provided by the research team on the Patient Screen, add a new patient on the Edit Patient Screen, add the Diabetes Family Responsibility Questionnaire on the Edit Patient Screen, create a survey access code to share with the patient.
  Groups: Physician Group
Behavioral: Front Desk Staff Intervention — On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen, choose patient Will Owens on the Visit Status Screen, add comments needs to be followed up regarding ketosis education in the comments for provider text box on the Visit Status Screen, add a goal for the patient log out of Goals-to-Guide application.
  Groups: Front Desk Staff
Behavioral: Nurse Intervention — On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen, choose patient Will Owens on the Visit Status screen, change HbA1C value to 10% on the Visit Status screen, change Nephropathy evaluation to Abnormal log out of Guide to Goals application.
  Groups: Nurses

SUMMARY:
The ultimate goal of this field trial is to systematically evaluate a novel care coordination tool for children with Type 2 Diabetes (T2D) in an office setting at Emory/Childrens Healthcare of Atlanta. The Guide to Goals (GTG) application was designed and developed at Georgia Institute of Technology with the aim of providing evidence-based information in a timely manner to all the stakeholders involved in the care of a T2D patient during an office visit

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the user interface of GTG for ease-of-use. By observing and analyzing actual user experience with the current version of the app investigators aim to learn about its shortcomings. Findings from this phase will be used to make GTG more user friendly. GTG is aimed at the following user groups: 1. Patients/caretakers 2. Font-desk staff 3. Nurses 4. Certified Diabetes Educators 5. Physicians In this phase, two participants will be recruited from each of the five user groups for a one-hour usability testing session during which time they will be subjected to the following: A. Introduction to study team and session procedures with the help of a physical consent form (15 minutes) B. Perform a set of tasks on the GTG application (15 minutes) C. Post task interview with study team (15 minutes) D. Fill out post-interview questionnaire (15 minutes) The specific set of tasks that each participants will perform during the usability testing session will be:

1. Front Desk Staff: On the Provider Login Screen, log in using the username and password provided by the research team on the Patient Screen, add a new patient on the Edit Patient Screen, add the Diabetes Family Responsibility Questionnaire on the Edit Patient Screen, create a survey access code to share with the patient.
2. Patient and/or Family Member: On the Patient Login Screen, log in using the last name and session ID provided by the research team on the Surveys Screen, click on a pending survey when the survey opens, respond to the survey submit the survey log out of the Guide-Goals Application.
3. Nurse: On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen, choose patient Will Owens on the Visit Status screen, change HbA1C value to 10% on the Visit Status screen, change Nephropathy evaluation to Abnormal log out of Guide to Goals application.
4. Certified Diabetes Educator: On the Provider Login Screen, log in using the participant's username and password provided by the research team on the Patients Screen, choose patient Will Owens on the Visit Status Screen, add comments needs to be followed up regarding ketosis education in the comments for provider text box on the Visit Status Screen, add a goal for the patient log out of Goals-to-Guide application.
5. Physician: On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen, choose patient Will Owens on the Visit Status Screen review planning and accountability sections for errors on the Visit Status Screen, add a goal for the patient log out of Goals- to-Guide application.

ELIGIBILITY:
Inclusion Criteria:

* Existing patients of Children's Healthcare of Atlanta (CHOA) with Type 2 Diabetes that are 12 or older at the time of participation or caretakers of existing patients of CHOA with Type 2 Diabetes
* Front desk staff
* Nurses at CHOA
* Certified Diabetes Educators at CHOA
* Physicians working at CHOA
* Participants must also be fluent in English, either as a first or secondary language, as the Guide-To-Goals app is in English.

Exclusion Criteria:

* Individuals that are using a care coordination tool other than GTG to translate ADA clinical standards of care for children with T2D during the study period will be excluded from this study in order to avoid confounding factors. Examples of care coordination tools include products that have the capabilities to send and receive electronic messages to the care team, receive and discuss care plans, and create and share health logs.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals participating in the usability testing session must be one the following: 1. Existing patients of Children's Healthcare of Atlanta (CHOA) with Type 2 Diabetes that are 12 or older at the time of participation or caretakers of existing patients of CHOA with Type 2 Diabetes 2. Front desk staff 3. Nurses at CHOA 4. Certified Diabetes Educators at CHOA 5. Physicians working at CHOA Participants must also be fluent in English, either as a first or secondary language, as the Guide-To-Goals app is in English.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiten Chhabra, MD, MS, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Children's Helathcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White NH, Sun W, Cleary PA, Tamborlane WV, Danis RP, Hainsworth DP, Davis MD; DCCT-EDIC Research Group. Effect of prior intensive therapy in type 1 diabetes on 10-year progression of retinopathy in the DCCT/EDIC: comparison of adults and adolescents. Diabetes. 2010 May;59(5):1244-53. doi: 10.2337/db09-1216. Epub 2010 Feb 11. PMID 20150283
- [Background] Kim H, Elmi A, Henderson CL, Cogen FR, Kaplowitz PB. Characteristics of children with type 1 diabetes and persistent suboptimal glycemic control. J Clin Res Pediatr Endocrinol. 2012 Jun;4(2):82-8. doi: 10.4274/jcrpe.663. PMID 22672865
- [Background] Silverstein J, Klingensmith G, Copeland K, Plotnick L, Kaufman F, Laffel L, Deeb L, Grey M, Anderson B, Holzmeister LA, Clark N; American Diabetes Association. Care of children and adolescents with type 1 diabetes: a statement of the American Diabetes Association. Diabetes Care. 2005 Jan;28(1):186-212. doi: 10.2337/diacare.28.1.186. No abstract available. PMID 15616254
- [Background] Bell RA, Mayer-Davis EJ, Beyer JW, D'Agostino RB Jr, Lawrence JM, Linder B, Liu LL, Marcovina SM, Rodriguez BL, Williams D, Dabelea D; SEARCH for Diabetes in Youth Study Group. Diabetes in non-Hispanic white youth: prevalence, incidence, and clinical characteristics: the SEARCH for Diabetes in Youth Study. Diabetes Care. 2009 Mar;32 Suppl 2(Suppl 2):S102-11. doi: 10.2337/dc09-S202. PMID 19246575
- [Background] Lawrence JM, Mayer-Davis EJ, Reynolds K, Beyer J, Pettitt DJ, D'Agostino RB Jr, Marcovina SM, Imperatore G, Hamman RF; SEARCH for Diabetes in Youth Study Group. Diabetes in Hispanic American youth: prevalence, incidence, demographics, and clinical characteristics: the SEARCH for Diabetes in Youth Study. Diabetes Care. 2009 Mar;32 Suppl 2(Suppl 2):S123-32. doi: 10.2337/dc09-S204. PMID 19246577
- [Background] Mayer-Davis EJ, Beyer J, Bell RA, Dabelea D, D'Agostino R Jr, Imperatore G, Lawrence JM, Liese AD, Liu L, Marcovina S, Rodriguez B; SEARCH for Diabetes in Youth Study Group. Diabetes in African American youth: prevalence, incidence, and clinical characteristics: the SEARCH for Diabetes in Youth Study. Diabetes Care. 2009 Mar;32 Suppl 2(Suppl 2):S112-22. doi: 10.2337/dc09-S203. PMID 19246576
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group; Nathan DM, Zinman B, Cleary PA, Backlund JY, Genuth S, Miller R, Orchard TJ. Modern-day clinical course of type 1 diabetes mellitus after 30 years' duration: the diabetes control and complications trial/epidemiology of diabetes interventions and complications and Pittsburgh epidemiology of diabetes complications experience (1983-2005). Arch Intern Med. 2009 Jul 27;169(14):1307-16. doi: 10.1001/archinternmed.2009.193. PMID 19636033
- [Background] Secrest AM, Becker DJ, Kelsey SF, Laporte RE, Orchard TJ. Cause-specific mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes. Diabetes. 2010 Dec;59(12):3216-22. doi: 10.2337/db10-0862. Epub 2010 Aug 25. PMID 20739685
- [Background] Wood JR, Miller KM, Maahs DM, Beck RW, DiMeglio LA, Libman IM, Quinn M, Tamborlane WV, Woerner SE; T1D Exchange Clinic Network. Most youth with type 1 diabetes in the T1D Exchange Clinic Registry do not meet American Diabetes Association or International Society for Pediatric and Adolescent Diabetes clinical guidelines. Diabetes Care. 2013 Jul;36(7):2035-7. doi: 10.2337/dc12-1959. Epub 2013 Jan 22. PMID 23340893
- [Background] Fogel NR, Weissberg-Benchell J. Preventing poor psychological and health outcomes in pediatric type 1 diabetes. Curr Diab Rep. 2010 Dec;10(6):436-43. doi: 10.1007/s11892-010-0145-z. PMID 20835901
- [Background] Bernstein CM, Stockwell MS, Gallagher MP, Rosenthal SL, Soren K. Mental health issues in adolescents and young adults with type 1 diabetes: prevalence and impact on glycemic control. Clin Pediatr (Phila). 2013 Jan;52(1):10-5. doi: 10.1177/0009922812459950. Epub 2012 Sep 17. PMID 22988007
- [Background] American Diabetes Association. Standards of medical care in diabetes--2013. Diabetes Care. 2013 Jan;36 Suppl 1(Suppl 1):S11-66. doi: 10.2337/dc13-S011. No abstract available. PMID 23264422
- [Background] Coleman K, Austin BT, Brach C, Wagner EH. Evidence on the Chronic Care Model in the new millennium. Health Aff (Millwood). 2009 Jan-Feb;28(1):75-85. doi: 10.1377/hlthaff.28.1.75. PMID 19124857
- [Background] Alliance CC. Chronic Care Management - Five More Chronics. In: Outcomes Guidelines Report. Washington, D.C.; 2010:55-118.
- [Background] Austin S, Senecal C, Guay F, Nouwen A. Effects of gender, age, and diabetes duration on dietary self-care in adolescents with type 1 diabetes: a Self-Determination Theory perspective. J Health Psychol. 2011 Sep;16(6):917-28. doi: 10.1177/1359105310396392. Epub 2011 Mar 23. PMID 21430132
- [Background] Whittemore R, Jaser S, Guo J, Grey M. A conceptual model of childhood adaptation to type 1 diabetes. Nurs Outlook. 2010 Sep-Oct;58(5):242-51. doi: 10.1016/j.outlook.2010.05.001. PMID 20934079
- [Background] Botello-Harbaum M, Nansel T, Haynie DL, Iannotti RJ, Simons-Morton B. Responsive parenting is associated with improved type 1 diabetes-related quality of life. Child Care Health Dev. 2008 Sep;34(5):675-81. doi: 10.1111/j.1365-2214.2008.00855.x. PMID 18796059
- [Background] Armstrong B, Mackey ER, Streisand R. Parenting behavior, child functioning, and health behaviors in preadolescents with type 1 diabetes. J Pediatr Psychol. 2011 Oct;36(9):1052-61. doi: 10.1093/jpepsy/jsr039. Epub 2011 Aug 9. PMID 21828111
- [Background] Wang YC, Stewart S, Tuli E, White P. Improved glycemic control in adolescents with type 1 diabetes mellitus who attend diabetes camp. Pediatr Diabetes. 2008 Feb;9(1):29-34. doi: 10.1111/j.1399-5448.2007.00285.x. PMID 18211634
- [Background] Iannotti RJ, Schneider S, Nansel TR, Haynie DL, Plotnick LP, Clark LM, Sobel DO, Simons-Morton B. Self-efficacy, outcome expectations, and diabetes self-management in adolescents with type 1 diabetes. J Dev Behav Pediatr. 2006 Apr;27(2):98-105. doi: 10.1097/00004703-200604000-00003. PMID 16682872
- [Background] Nouwen A, Urquhart Law G, Hussain S, McGovern S, Napier H. Comparison of the role of self-efficacy and illness representations in relation to dietary self-care and diabetes distress in adolescents with type 1 diabetes. Psychol Health. 2009 Nov;24(9):1071-84. doi: 10.1080/08870440802254597. PMID 20205046
- [Background] Robinson EM, Iannotti RJ, Schneider S, Nansel TR, Haynie DL, Sobel DO. Parenting goals: predictors of parent involvement in disease management of children with type 1 diabetes. J Child Health Care. 2011 Sep;15(3):199-209. doi: 10.1177/1367493511406567. PMID 21917595
- [Background] Modi AC, Pai AL, Hommel KA, Hood KK, Cortina S, Hilliard ME, Guilfoyle SM, Gray WN, Drotar D. Pediatric self-management: a framework for research, practice, and policy. Pediatrics. 2012 Feb;129(2):e473-85. doi: 10.1542/peds.2011-1635. Epub 2012 Jan 4. PMID 22218838
- [Background] Holtz B, Lauckner C. Diabetes management via mobile phones: a systematic review. Telemed J E Health. 2012 Apr;18(3):175-84. doi: 10.1089/tmj.2011.0119. Epub 2012 Feb 22. PMID 22356525
- [Background] Mulvaney SA, Ritterband LM, Bosslet L. Mobile intervention design in diabetes: review and recommendations. Curr Diab Rep. 2011 Dec;11(6):486-93. doi: 10.1007/s11892-011-0230-y. PMID 21960031
- [Background] Eng DS, Lee JM. The promise and peril of mobile health applications for diabetes and endocrinology. Pediatr Diabetes. 2013 Jun;14(4):231-8. doi: 10.1111/pedi.12034. Epub 2013 Apr 30. PMID 23627878
- [Background] El-Gayar O, Timsina P, Nawar N, Eid W. A systematic review of IT for diabetes self-management: are we there yet? Int J Med Inform. 2013 Aug;82(8):637-52. doi: 10.1016/j.ijmedinf.2013.05.006. Epub 2013 Jun 21. PMID 23792137
- [Background] Waitzfelder B, Pihoker C, Klingensmith G, Case D, Anderson A, Bell RA, Lawrence JM, Mayer-Davis EJ, Imperatore G, Standiford D, Rodriguez BL, Dabelea D, Seid M; SEARCH for Diabetes in Youth Study Group. Adherence to guidelines for youths with diabetes mellitus. Pediatrics. 2011 Sep;128(3):531-8. doi: 10.1542/peds.2010-3641. Epub 2011 Aug 22. PMID 21859914
- [Background] Eijkenaar F, Emmert M, Scheppach M, Schoffski O. Effects of pay for performance in health care: a systematic review of systematic reviews. Health Policy. 2013 May;110(2-3):115-30. doi: 10.1016/j.healthpol.2013.01.008. Epub 2013 Feb 4. PMID 23380190
- [Background] Berman B, Pracilio VP, Crawford A, Behm WR, Jacoby R, Nash DB, Goldfarb NI. Implementing the physician quality reporting system in an academic multispecialty group practice: lessons learned and policy implications. Am J Med Qual. 2013 Nov-Dec;28(6):464-71. doi: 10.1177/1062860613476733. Epub 2013 Mar 12. PMID 23482676
- [Background] Kovacs M. The Children's Depression, Inventory (CDI). Psychopharmacol Bull. 1985;21(4):995-8. No abstract available. PMID 4089116
- [Background] Markowitz JT, Butler DA, Volkening LK, Antisdel JE, Anderson BJ, Laffel LM. Brief screening tool for disordered eating in diabetes: internal consistency and external validity in a contemporary sample of pediatric patients with type 1 diabetes. Diabetes Care. 2010 Mar;33(3):495-500. doi: 10.2337/dc09-1890. Epub 2009 Dec 23. PMID 20032278
- [Background] Helgeson VS, Reynolds KA, Siminerio L, Escobar O, Becker D. Parent and adolescent distribution of responsibility for diabetes self-care: links to health outcomes. J Pediatr Psychol. 2008 Jun;33(5):497-508. doi: 10.1093/jpepsy/jsm081. Epub 2007 Sep 10. PMID 17848390
- See also: Link to the coordination tool application — http://G2g.gatech.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in the following sequence of events: 1. Members of Dr. Andrew Muir's staff at CHOA described the study to potential participants during regular office visits. 2. Individuals interested in participating in the study then schedules a time to meet with a member of the study team at CHOA and consented to be part of the study.
Period: Overall Study
Arm/Group | Patients/Caretakers Group | Certified Diabetes Educators Group | Physician Group | Front Desk Staff | Nurses
Started | 1 | 1 | 0 (Not Completed) | 2 | 2
Completed | 1 | 1 | 0 (Not Completed) | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study team could not recruit 2 physicians due to the limitations imposed by COVID-19 during the recruitment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients/Caretakers Group | Certified Diabetes Educators Group | Physician Group | Front Desk Staff | Nurses | Total
Number analyzed (Participants) | 1 | 1 | 0 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 2 | 2 | 6
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 1 | 4
  Male | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 1 | 1 | 0 | 1 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Participant Task Completion Rate for Usability Testing Session
Description: Number of participants that complete all the tasks assigned to them during the intervention (usability testing session).
Time Frame: 1 month
Population: Recruitment incomplete due to COVID-19
Measure: Count of Participants; unit: Participants
Arm/Group | Patients/Caretakers Group | Certified Diabetes Educators Group | Physician Group | Front Desk Staff | Nurses
Number analyzed (Participants) | 1 | 1 | 0 | 2 | 2
Participants | 1 | 1 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 1 Month
Description: No participants were enrolled in the Physician Arm due to COVID-19
Arm/Group | Patients/Caretakers Group | Certified Diabetes Educators Group | Physician Group | Front Desk Staff | Nurses
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (5):
  • Study Protocol (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03926598/Prot_003.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03926598/SAP_004.pdf
  • Informed Consent Form: Adult Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03926598/ICF_000.pdf
  • Informed Consent Form: Minor Assent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03926598/ICF_001.pdf
  • Informed Consent Form: Parental Permission Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03926598/ICF_002.pdf